CLINICAL TRIAL: NCT04475588
Title: A Multi-Centre, Open Label, Two Arm Randomized, Phase 2 Trial to Study the Efficacy and Safety of Itolizumab in COVID-19 Complications
Brief Title: Efficacy and Safety of Itolizumab in COVID-19 Complications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biocon Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITOLI-C19-02-I-00
Record Dates: First submitted 2020-07-16; First posted 2020-07-17 (Actual); Results first posted 2021-05-20 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Acute Respiratory Distress Syndrome; Cytokine Release Syndrome; Covid19
MeSH Terms: conditions — Respiratory Distress Syndrome; Cytokine Release Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Itolizumab + BSC (Experimental)
  Interventions: Drug: Itolizumab IV infusion; Drug: Best supportive care (BSC)
- Arm B - Best supportive care (BSC) (Active Comparator)
  Interventions: Drug: Best supportive care (BSC)

INTERVENTIONS:
Drug: Itolizumab IV infusion — First dose of 1.6 mg/kg dose iv infusion, , investigator discretion to continue with 1.6 mg/kg dose every 2 weeks or 0.8 mg/kg weekly regimen up to 4 weeks.
  BSC: similar to Arm B
  Arms: Arm A - Itolizumab + BSC
Drug: Best supportive care (BSC) — Best supportive care (BSC) included drugs like antivirals, antibiotics, Hydroxychloroquine, oxygen therapy, LMWH, Steroids, Vitamins and Zinc

SUMMARY:
Randomized, Parallel Group, Active Controlled Trial

DETAILED DESCRIPTION:
This is a Multi-Centric, Open label, Two Arm Randomized, Phase 2 Study.

All eligible patients entering into the study will be randomized in 2:1 ratio to receive the treatment A (Best supportive care + Itolizumab) / B (Best supportive care) respectively. Each patient will undergo the treatment based on their assigned treatment for a month along with battery of tests that includes, but not limited to, cytokines and chemokine, along with recording of TLC; DLC, ANC, ALC; Platelet count; S. creatinine; T.Bilirubin; morning Vitals -pulse, BP, RR; Temperature, PaO2/FiO2, MAP, GCS.

As Itolizumab is an investigational drug, the benefit to COVID-19 patients experiencing complications such as Cytokine Release Syndrome is not known. However, findings from this study may be beneficial to the society at a large at the National and International Level.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female adults above 18 years (not tested in children yet)
2. Informed consent for participation in the study
3. Virological diagnosis of SARS-CoV2 infection (PCR)
4. Hospitalized due to clinical/instrumental diagnosis of COVID-19 infection
5. Oxygen saturation at rest in ambient air ≤94%
6. Patients who are in moderate to severe ARDS as defined by PaO2/Fio2 ratio of < 200

Key Exclusion Criteria:

1. Known severe allergic reactions to monoclonal antibodies
2. Active tuberculosis (TB) infection
3. History of inadequately treated tuberculosis or latent tuberculosis
4. In the opinion of the investigator,progression to death is highly probable, irrespective of the provision of treatments
5. Have received oral anti-rejection or immune-suppressive drugs within the past 6 months
6. Participating in other drug clinical trials (participation in COVID-19 anti-viral trials may be permitted if approved by Medical Monitor)
7. Pregnant or breastfeeding, or positive pregnancy test in a pre-dose examination
8. Patients with known history of Hepatitis B, Hepatitis C or HIV
9. Absolute Neutrophils count (ANC) <1000 / mm3
10. Platelets <50,000 / mm3
11. Absolute Lymphocyte count (ALC): <500/mm3

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- India (4):
  - Topiwala National Medical College & B. Y. L. Nair Charitable Hospital,, Mumbai
  - Seth GS Medical College and KEM Hospital, Mumbai
  - MAMC medical college and Lok Nayak Jai Prakash Narayan Hospital hospital, New Delhi
  - All India Institute Of Medical Sciences, New Delhi

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Itolizumab + BSC: Itolizumab IV infusion Itolizumab IV infusion: First dose of 1.6 mg/kg dose iv infusion, , investigator discretion to continue with 1.6 mg/kg dose every 2 weeks or 0.8 mg/kg weekly regimen up to 4 weeks.
  BSC: similar to Arm B Drug: Best supportive care (BSC) included drugs like antivirals, antibiotics, Hydroxychloroquine, oxygen therapy, LMWH, Steroids, Vitamins and Zinc
- Arm B - Best Supportive Care (BSC): Best supportive care (BSC) included drugs like antivirals, antibiotics, Hydroxychloroquine, oxygen therapy, LMWH, Steroids, Vitamins and Zinc
Period: Overall Study
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Started | 22 (Stated in protocol apriori, patient not completing 1st infusion were not evaluable & were replaced.) | 10
Completed | 20 | 10
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A - Itolizumab + BSC: IItolizumab IV infusion Itolizumab IV infusion: First dose of 1.6 mg/kg dose iv infusion, , investigator discretion to continue with 1.6 mg/kg dose every 2 weeks or 0.8 mg/kg weekly regimen up to 4 weeks.
  BSC: similar to Arm B Drug: Best supportive care (BSC) included drugs like antivirals, antibiotics, Hydroxychloroquine, oxygen therapy, LMWH, Steroids, Vitamins and Zinc
- Total: Total of all reporting groups
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC) | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.55 (12.49) | 48.30 (14.62) | 49.13 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 19 | 7 | 26
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 20 | 10 | 30
Region of Enrollment [Number; unit: participants]
  India | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: One-month Mortality Rate Between the Two Arms
Description: 1-month mortality is defined as the proportion of patients who met fatal outcome event by Day 30
Time Frame: One-month
Measure: Number; unit: participants
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 20 | 10
participants | 0 | 3

2. Primary Outcome: Lung Function Assessment - Proportion of the Patients With Stable or Improved SpO2 Without Increasing FiO2
Description: Stable SpO2: Defined as number of patients with absence of increase in FiO2 to maintain SpO2 ≥ 92% Improvement of SpO2: Defined as number of patients with decrease in FiO2 to maintain SpO2 > 92%
Time Frame: Day 7, Day 14, Day 21 & Day 30
Population: Patients improved/ weaned off O2, the observation was carried forward
Measure: Number; unit: participants
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 20 | 10
participants
  Day 7 | 17 | 5
  Day 14 | 19 | 7
  Day 21 | 20 | 7
  Day 30/EOS | 20 | 7

3. Primary Outcome: Endo-tracheal Intubation/Invasive Mechanical Ventilation (IMV)
Description: Number of patients needing Intubation/IMV post treatment
Time Frame: Day 30
Measure: Number; unit: participants
Groups:
- Arm A - Itolizumab + BSC: Itolizumab IV infusion Itolizumab IV infusion: First dose of 1.6 mg/kg dose iv infusion, , investigator discretion to continue with 1.6 mg/kg dose every 2 weeks or 0.8 mg/kg weekly regimen up to 4 weeks.
  BSC: similar to Arm B Drug: Best supportive care (BSC) included drugs like antivirals, antibiotics, Hydroxychloroquine, oxygen therapy, LMWH,Steroids,Vitamins and Zinc
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 20 | 10
participants | 0 | 2

4. Primary Outcome: Reduction in Proportion of Patients on Non-invasive Ventilation
Description: Reduction in proportion of Patients on Non-invasive Ventilation: defined as number of patient improved and shifted to Face mask, Nasal cannula, non-rebreather mask or off oxygen over time
Time Frame: Baseline (Day 1), Day 7, Day 14 Day 21 & Day 30
Measure: Number; unit: participants
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 20 | 10
participants
  Baseline (Day 1) | 5 | 4
  Day 7 | 0 | 0
  Day 14 | 5 | 1
  Day 21 | 5 | 1
  Day 30/EOS | 5 | 1

5. Primary Outcome: Lung Function Assessment - Proportion of Patients With Stable PaO2 Without Increasing FiO2
Description: Stable PaO2: Defined as number of patients with up to 10% change in PaO2/FiO2 ratio from baseline.
  Improvement of PaO2: Defined as number of patients with > 10% improvement in PaO2/FiO2 ratio from baseline (including patients weaned off oxygen).
Time Frame: Day 7, Day14, Day 21 & Day30
Population: Patients improved/ weaned off O2, the observation was carried forward.
Measure: Number; unit: participants
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 20 | 10
participants
  Day 7 | 18 | 6
  Day 14 | 19 | 7
  Day 21 | 20 | 7
  Day 30/EOS | 20 | 7

6. Primary Outcome: Reduction in Proportion of Patients- Invasive Mechanical Ventilation
Description: Patient improved from invasive ventilation over time from baseline.
Time Frame: Day7, Day14, Day21 & Day 30
Population: There were no patients on invasive mechanical ventilation at baseline
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Reduction in Proportion of Patients-High Flow Nasal Oxygen
Description: Patient improved from High Flow Nasal Oxygen over time from baseline.
Time Frame: Day7 ,Day 14 ,Day 21, Day 30
Population: There were no patients on High Flow Nasal Oxygen at baseline
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Mean Change From Baseline in Ferritin
Description: Mean Change from Baseline in Ferritin
Time Frame: Day 7, Day 14, Day 21 & Day 30
Population: only "observed values" were used.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 20 | 10
ng/mL
  Day 7: number analyzed (Participants) | 18 | 7
  Day 7 | -117.8 (1477.0) | -87.05 (140.99)
  Day 14: number analyzed (Participants) | 15 | 5
  Day 14 | -713.9 (693.68) | -209.6 (177.33)
  Day 21: number analyzed (Participants) | 11 | 3
  Day 21 | -780.9 (630.61) | 4238 (8319.0)
  Day 30/EOS: number analyzed (Participants) | 3 | 2
  Day 30/EOS | -479.3 (620.95) | -234.4 (405.67)

9. Primary Outcome: Mean Change From Baseline in LDH
Description: Mean Change from Baseline in LDH
Time Frame: Day 7, Day14, Day 21 and Day 30.
Population: Only "observed values" were used.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 20 | 10
U/L
  Day 7: number analyzed (Participants) | 18 | 7
  Day 7 | -134 (174.67) | -44.29 (176.85)
  Day 14: number analyzed (Participants) | 15 | 5
  Day 14 | -195.8 (291.94) | -195.2 (119.93)
  Day 21: number analyzed (Participants) | 11 | 3
  Day 21 | -308.1 (202.76) | 155.3 (736.47)
  Day 30/EOS: number analyzed (Participants) | 3 | 2
  Day 30/EOS | -212.7 (188.48) | -97 (89.1)

10. Primary Outcome: Mean Change From Baseline in CRP (C-reactive Protein)
Description: Mean Change from Baseline in CRP
Time Frame: Day 7, Day 14, Day 21 & Day 30
Population: Only "observed values" were used.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 20 | 10
mg/L
  Day 7: number analyzed (Participants) | 18 | 8
  Day 7 | -61.69 (81.86) | -103.6 (87.48)
  Day 14: number analyzed (Participants) | 16 | 5
  Day 14 | -81.65 (74.71) | -107.2 (104.66)
  Day 21: number analyzed (Participants) | 11 | 3
  Day 21 | -90.99 (81.97) | -127.5 (124.04)
  Day 30/EOS: number analyzed (Participants) | 3 | 2
  Day 30/EOS | -103.2 (100.53) | -127.6 (59.68)

11. Primary Outcome: Mean Change From Baseline D-Dimer
Time Frame: Day 7, Day 14, Day 21 & Day 30
Population: Only "observed values" were used.
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 20 | 10
µg/ml
  Day 7: number analyzed (Participants) | 18 | 7
  Day 7 | -1.43 (6.31) | 2.30 (6.67)
  Day 14: number analyzed (Participants) | 12 | 4
  Day 14 | -0.45 (6.39) | -0.68 (0.79)
  Day 21: number analyzed (Participants) | 11 | 2
  Day 21 | -4.35 (6.13) | 8.54 (14.40)
  Day 30: number analyzed (Participants) | 3 | 2
  Day 30 | -2.63 (2.43) | -0.35 (0.08)

12. Secondary Outcome: Mean Change From Baseline of Absolute Lymphocyte Count
Description: Mean change From baseline in Lymphocyte count
Time Frame: day 7, day 14 ,day 21 & day 30
Population: Only "observed values" were used.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 20 | 10
cells/mm^3
  Day 7: number analyzed (Participants) | 20 | 8
  Day 7 | 119.95 (478.63) | 45.88 (762.37)
  Day 14: number analyzed (Participants) | 16 | 5
  Day 14 | 421.25 (569.71) | 142.60 (731.94)
  Day 21: number analyzed (Participants) | 11 | 3
  Day 21 | 701.55 (625.34) | 10.00 (930.16)
  Day 30/EOS: number analyzed (Participants) | 4 | 2
  Day 30/EOS | 719.75 (1004.0) | 85.00 (601.04)

13. Secondary Outcome: Biomarkers (IL-6, TNF-a)
Description: Mean values of Pre and Post 1st and 2nd dose are shown
Time Frame: Pre and Post 1st dose; Pre and Post 2nd dose
Population: Only "observed values" were used.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 18 | 10
pg/ml
  IL-6 (Pre 1st Dose) | 159.09 (293.0) | 162.16 (185.9)
  IL-6 (Post 1st Dose) | 42.98 (52.9) | 211.52 (297.2)
  IL-6 (Pre 2nd Dose): number analyzed (Participants) | 13 | 4
  IL-6 (Pre 2nd Dose) | 311.3 (660.4) | 310.4 (528.2)
  IL-6 (Post 2nd Dose): number analyzed (Participants) | 13 | 4
  IL-6 (Post 2nd Dose) | 91.0 (245.6) | 316.8 (373.7)
  TNF-a (Pre 1st Dose) | 43.64 (72.9) | 11.26 (13.6)
  TNF-a (Post 1st Dose) | 8.87 (12.3) | 39.19 (104.5)
  TNF-a (Pre 2nd Dose: number analyzed (Participants) | 13 | 4
  TNF-a (Pre 2nd Dose | 68.0 (109.5) | 107.8 (175.3)
  TNF-a (Post 2nd Dose): number analyzed (Participants) | 13 | 4
  TNF-a (Post 2nd Dose) | 50.1 (140.2) | 185.0 (275.8)

14. Secondary Outcome: Mean PaO2 (Partial Pressure of Oxygen) / FiO2 (Fraction of Inspired Oxygen, FiO2) Ratio (or P/F Ratio)
Description: Mean PaO2 (partial pressure of oxygen) / FiO2 (fraction of inspired oxygen, FiO2) ratio (or P/F ratio)
Time Frame: Baseline, Day 7, Day 14, Day 21 & Day 30
Population: Only "observed values" were used.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 20 | 10
Ratio
  Baseline/Day 1 | 126.57 (38.31) | 114.05 (30.93)
  Day 7: number analyzed (Participants) | 16 | 6
  Day 7 | 203.50 (95.51) | 184.53 (95.51)
  Day 14: number analyzed (Participants) | 14 | 5
  Day 14 | 283.43 (104.26) | 338.40 (42.57)
  Day 21: number analyzed (Participants) | 8 | 3
  Day 21 | 350.25 (70.36) | 398.33 (24.01)
  Day 30/EOS: number analyzed (Participants) | 3 | 0
  Day 30/EOS | 397.67 (15.63) |

15. Secondary Outcome: Number and Percentage of Patients With Radiological Response
Description: Number of patients with improved X ray/CT findings as compared to baseline or returned to normal in the last assessment
Time Frame: up to Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
Number analyzed (Participants) | 20 | 10
Participants | 9 | 1

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Arm A - Itolizumab + BSC | Arm B - Best Supportive Care (BSC)
All-Cause Mortality (participants affected / at risk) | 1/22 | 3/10
Serious Adverse Events (participants affected / at risk) | 3/22 | 3/10
Other Adverse Events (participants affected / at risk) | 18/22 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Itolizumab + BSC (N=22) | Arm B - Best Supportive Care (BSC) (N=10)
Pericardial effusion due to underlying hypothyroidism (Cardiac disorders) | 1 (1) | 0 (0) — Unrelated event in Arm A
Anaphylactic reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Related event in Arm A
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) — Outcome death, in Arm B
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Outcome was death, in Arm B
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Patient had Infusion Reaction, did not complete initial dose. Event resolved same day. Per protocol, patient not completing first infusion were not evaluable & were replaced. Patient recovered & was discharged 2-wks later.
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Itolizumab + BSC (N=22) | Arm B - Best Supportive Care (BSC) (N=10)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 5 (6) | 0 (0) — 1 Pt. had chills did not complete initial dose. Event resolved same day. Per protocol pt. not completing 1 dose were not evaluable & replaced. Pt had COVID19 complications, death 9 days later, deemed not related to drug. Stated in all cause mortality
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 11 (11) | 2 (2)
Non-high-density lipoprotein cholesterol increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to current pandemic situation few datapoints not available for ptxs who got discharged earlier basis clinical status & bed shortage. As time to discharge was influenced by load on the hospital it was not an evaluable parameter after the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT04475588/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT04475588/SAP_001.pdf